CLINICAL TRIAL: NCT00973609
Title: Randomized Three Arm Phase III Trial on Induction Treatment With a Fluoropyrimidine-, Oxaliplatin- and Bevacizumab-based Chemotherapy for 24 Weeks Followed by Maintenance Treatment With a Fluoropyrimidine and Bevacizumab vs. Bevacizumab Alone vs. no Maintenance Treatment and Reinduction in Case of Progression for First-line Treatment of Patients With Metastatic Colorectal Cancer
Brief Title: Optimal Maintenance Therapy With Bevacizumab After Induction in Metastatic Colorectal Cancer (CRC)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: AIO-Studien-gGmbH (Other)
Collaborators: Roche Pharma AG (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: AIO-KRK-0207; ML21768; EudraCT-Nr.: 2008-007974-39
Record Dates: First submitted 2009-08-19; First posted 2009-09-09 (Estimated); Last update posted 2015-09-01 (Estimated); Status verified 2015-08

CONDITIONS: Colorectal Neoplasms
Keywords: metastatic colorectal cancer; Bevacizumab; Avastin®; phase 3; maintenance treatment; treatment pause; drug holiday; stage IV
MeSH Terms: conditions — Colorectal Neoplasms | interventions — Fluorouracil; Folic Acid; Capecitabine; Bevacizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Fluoropyrimidine + Bevacizumab (Active Comparator): Standard therapy
  Interventions: Drug: 5-Fluorouracil, Folic acid, Capecitabine; Bevacizumab
- Bevacizumab monotherapy (Experimental)
  Interventions: Drug: 5-Fluorouracil, Folic acid, Capecitabine; Bevacizumab
- No maintenance treatment (Experimental)
  Interventions: Drug: 5-Fluorouracil, Folic acid, Capecitabine; Bevacizumab

INTERVENTIONS:
Drug: 5-Fluorouracil, Folic acid, Capecitabine; Bevacizumab — Induction (and reinduction) treatment regimen for 24 weeks: Fluoropyrimidine, oxaliplatin and bevacizumab.
  Following induction treatment regimen (for maintenance treatment): No maintenance treatment.
  Arms: No maintenance treatment
Drug: 5-Fluorouracil, Folic acid, Capecitabine; Bevacizumab — Induction (and reinduction) treatment regimen for 24 weeks: Fluoropyrimidine, oxaliplatin and bevacizumab.
  Following induction treatment regimen (for maintenance treatment): Fluoropyrimidine + Bevacizumab.
  Arms: Fluoropyrimidine + Bevacizumab
Drug: 5-Fluorouracil, Folic acid, Capecitabine; Bevacizumab — Induction (and reinduction) treatment regimen for 24 weeks: Fluoropyrimidine, oxaliplatin and bevacizumab.
  Following induction treatment regimen (for maintenance treatment): Bevacizumab monotherapy.
  Arms: Bevacizumab monotherapy

SUMMARY:
Investigating the efficacy of maintenance and reinduction treatment or no treatment and watchful waiting in subjects with inoperable or irresectable and non-progressive metastatic colorectal cancer after first line induction treatment for 24 weeks with a fluoropyrimidine-, oxaliplatin- and bevacizumab-based chemotherapy.

The maintenance treatment with capecitabine or 5-FU/folinic acid and bevacizumab will be compared with a maintenance treatment with bevacizumab alone or no maintenance treatment. Reinduction treatment will be done in case of progression.

DETAILED DESCRIPTION:
Chemotherapy and bevacizumab represent a standard of care in treatment of metastatic colorectal cancer. Until now, continuation of chemotherapy - and bevacizumab - represents the standard of care in colorectal cancer treatment. However, since the OPTIMOX1 trial showed an equivalent duration of disease control for a de-escalation / maintenance / reintroduction strategy compared with a treatment until progression strategy for oxaliplatin-based chemotherapy, the question is whether this strategy might apply also to bevacizumab in combination with chemotherapy. Furthermore, with the introduction of bevacizumab, there are new options for a maintenance treatment which should be evaluated.

As the continuation of chemotherapy plus bevacizumab until disease progression has to be regarded as standard of care, the question is whether a de-escalation of treatment intensity or even withdrawal of treatment ("drug holiday") after a certain treatment period will not be inferior with respect to resulting time with tumor control, but allow patients a period with less toxicity and gain of quality of life.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed and inoperable or irresectable metastatic colorectal cancer (stage IV)
* Measurable lesion according to RECIST measured within 4 weeks prior to registration of the subject for the study
* Not allowed prior treatments:

  * Previous chemotherapy for metastatic disease (adjuvant therapy for non-metastasized disease is allowed if terminated more than 6 months ago and without recurrence within 6 months after the end of adjuvant treatment)
  * Prior radiation of indicator lesion(s), except for documented progression during radiation and termination of radiotherapy at least 4 weeks prior to entry into the study
* 18 and over
* ECOG 0-2
* Prior and concomitant associated diseases:

  * No past or current history of malignancies except for the indication under this study and curatively treated:

    * Basal and squamous cell carcinoma of the skin
    * in situ carcinoma of the cervix
    * Other malignant disease without recurrence after at least 5 years of follow-up
  * No severe internal disease (insufficiently treated or uncontrolled arterial hypertension, haemoptoe, New York Heart Association (NYHA) grade II or greater congestive heart failure, symptomatic coronary heart disease, myocardial infarction (= < 12 months prior to inclusion), serious cardiac arrhythmia requiring medication, peripheral arterial occlusive disease stage II or greater, uncontrolled severe disease)
  * No history or evidence upon physical examination of CNS disease unless adequately treated (e.g., primary brain tumour, seizure not controlled with standard medical therapy, brain metastases or history of stroke).
  * No pre-existing neuropathy > = grade 1 (NCI CTCAE), except for loss of tendon reflex as the only symptom
  * No interstitial pneumonia or symptomatic fibrosis of the lung
  * No allogenic transplantation requiring immuno-suppressive therapy
  * No severe non-healing wounds, ulcers or bone fractions.
  * No thrombosis or severe bleeding within 6 months prior to entry into the study (except for bleeding of the tumor before its surgical resection) and no evidence of bleeding diathesis or coagulopathy.
* Laboratory requirements - within 7 days prior to enrollment:

  * Neutrophil count > = 1,500/μl
  * Platelets > = 100,000/μl
  * Hb > = 9g/dl dL (may be transfused to maintain or exceed this level)
  * Serum creatinine clearance > 50ml/min (Cockroft/Gault)
  * Serum total bilirubin: = < 1.5 x UNL
  * AST and ALT = < 2.5 x UNL; = < 5 x UNL in subjects with documented liver metastases
* Patients not receiving therapeutic anticoagulation must have an INR < 1.5 ULN and aPTT < 1.5 ULN within 7 days prior to registration. The use of full dose anticoagulants is allowed as long as the INR or aPTT is within therapeutic limits (according to the medical standard in the institution) and the patient has been on a stable dose for anticoagulants for at least two weeks at the time of registration.
* Laboratory requirements in fertile women, within 2 days prior to treatment: Negative serum pregnancy test
* Other medication:

  * No concomitant therapy with certain anti-viral medicines (sorivudine and brivudine or analogue compounds).
  * No continuous medication with ASS > 325 mg or NSAIDs, known to inhibit platelet function.
* Other:

  * No major surgical procedure, open biopsy, nor significant traumatic injury within 28 days prior to study treatment start, nor anticipation of the need for major surgical procedure during the course of the study except for surgery for colorectal cancer with curative intent and central venous line placement for chemotherapy administration, which must be inserted at least 2 days prior to treatment start.
  * No pregnancy or breastfeeding women.
  * No women of child-bearing potential with positive or missing pregnancy test at study entry; post-menopausal women must have been amenorrheic for at least 12 months to be considered of non-child-bearing potential.
  * No sexually active men or women of childbearing potential not willing to use effective means of contraception (intrauterine contraceptive device, implants, injectables, sexual abstinence or vasectomised partner).
  * No subjects with known allergy to the used study drugs or to any of its excipients.
  * No known DPD deficiency.
  * No proteinuria (>1+); if dipstick test of urine exceeds 1+, proteinuria has to be below 1g protein in 24 hours urine.
  * No concomitant treatment with preparations of St. John's wort.
  * No currently or recent (within the 28 days prior to starting study treatment) treatment of another investigational drug or participation in another investigational study.
  * No known grade III/IV allergic reaction against monoclonal antibodies.
  * Absence of any psychological, familial, sociological or geographical condition potentially hampering compliance with the study protocol and follow-up schedule; those conditions should be discussed with the subject before registration in the trial.
  * Before subject registration, written informed consent must be given according to ICH/GCP, and national/local regulations. The subject must be competent to comprehend, sign, and date an IEC-approved informed consent form.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 853 (Actual)
Dates: Start 2009-08; Primary Completion 2014-12 (Actual); Study Completion 2015-08 (Actual)

PRIMARY OUTCOMES:
Time to failure of maintenance and reinduction treatment strategy measured from randomization | From randomization until second progression after reinduction treatment

SECONDARY OUTCOMES:
TFS, Toxicity, QoL, PFS 1, PFS 2, ORR (first induction), ORR (reind. treatm.), Treatment free interval/duration of maintenance therapy, second. Resection rate, Reasons for discontinuation, OS, Translational research. | From enrollment until second progression after reinduction treatment

CONTACTS AND LOCATIONS:
Overall Officials: Susanna Hegewisch-Becker, Prof. Dr., Principal Investigator — Onkologische Schwerpunktpraxis Eppendorf 20249 Hamburg Germany
Locations (1):
- AIO-Studien gGmbH, Berlin, State of Berlin, Germany

REFERENCES:
- [Derived] Lueong SS, Herbst A, Liffers ST, Bielefeld N, Horn PA, Tannapfel A, Reinacher-Schick A, Hinke A, Hegewisch-Becker S, Kolligs FT, Siveke JT. Serial Circulating Tumor DNA Mutational Status in Patients with KRAS-Mutant Metastatic Colorectal Cancer from the Phase 3 AIO KRK0207 Trial. Clin Chem. 2020 Dec 1;66(12):1510-1520. doi: 10.1093/clinchem/hvaa223. PMID 33257977
- [Derived] Hegewisch-Becker S, Nopel-Dunnebacke S, Hinke A, Graeven U, Reinacher-Schick A, Hertel J, Lerchenmuller CA, Killing B, Depenbusch R, Al-Batran SE, Lange T, Dietrich G, Tannapfel A, Arnold D. Impact of primary tumour location and RAS/BRAF mutational status in metastatic colorectal cancer treated with first-line regimens containing oxaliplatin and bevacizumab: Prognostic factors from the AIO KRK0207 first-line and maintenance therapy trial. Eur J Cancer. 2018 Sep;101:105-113. doi: 10.1016/j.ejca.2018.06.015. Epub 2018 Jul 20. PMID 30036739
- [Derived] Quidde J, Hegewisch-Becker S, Graeven U, Lerchenmuller CA, Killing B, Depenbusch R, Steffens CC, Lange T, Dietrich G, Stoehlmacher J, Reinacher A, Tannapfel A, Trarbach T, Marschner N, Schmoll HJ, Hinke A, Al-Batran SE, Arnold D. Quality of life assessment in patients with metastatic colorectal cancer receiving maintenance therapy after first-line induction treatment: a preplanned analysis of the phase III AIO KRK 0207 trial. Ann Oncol. 2016 Dec;27(12):2203-2210. doi: 10.1093/annonc/mdw425. Epub 2016 Oct 17. PMID 27753609
- [Derived] Hegewisch-Becker S, Graeven U, Lerchenmuller CA, Killing B, Depenbusch R, Steffens CC, Al-Batran SE, Lange T, Dietrich G, Stoehlmacher J, Tannapfel A, Reinacher-Schick A, Quidde J, Trarbach T, Hinke A, Schmoll HJ, Arnold D. Maintenance strategies after first-line oxaliplatin plus fluoropyrimidine plus bevacizumab for patients with metastatic colorectal cancer (AIO 0207): a randomised, non-inferiority, open-label, phase 3 trial. Lancet Oncol. 2015 Oct;16(13):1355-69. doi: 10.1016/S1470-2045(15)00042-X. Epub 2015 Sep 8. PMID 26361971
- See also: Related Info — http://www.aio-portal.de